CLINICAL TRIAL: NCT05281237
Title: Feasibility and Efficacy of the AveCure Flexible Microwave Ablation Probe for Peripheral Lung Nodule
Brief Title: Avecure Flexible Microwave Ablation Probe For Lung Nodules
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: MedWaves, Inc (Unknown); Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Jason A Beattie, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-412
Record Dates: First submitted 2022-02-16; First posted 2022-03-16 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Stage I - II Primary Lung Cancer; Stage I Lung Cancer; Stage II Lung Cancer; Lung Cancer Stage I; Lung Cancer Stage II; Lung Cancer
Keywords: Stage I - II primary lung cancer; Stage I Lung Cancer; Stage II Lung Cancer; Lung Cancer Stage I; Lung Cancer Stage II; Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- AVECURE FLEXIBLE MICROWAVE ABLATION PROBE FOR LUNG NODULES (Experimental): The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.
  * Ablation Procedure- MWA will be used to treat solitary pulmonary nodules up to 3cm.
  * CT scan will then be performed to evaluate the radiological changes 2 - 4 weeks after the ablation procedure.
  * Surgery will be performed to remove the lung nodule and the tissue will be evaluated by pathology.
  Interventions: Device: AveCure 16 Gauge Flexible Microwave Ablation Probe

INTERVENTIONS:
Device: AveCure 16 Gauge Flexible Microwave Ablation Probe — Microwave ablation of the solitary pulmonary nodule will be performed through a bronchoscopic approach using the AveCure Flexible Microwave Ablation Probe before surgery
  Other Names: Avecure

SUMMARY:
This research study to determine the effectiveness of the AveCure Flexible Microwave Ablation Probe to destroy cancerous lung nodules up to 3 c m in size.

This research study involves microwave ablation (MWA)

DETAILED DESCRIPTION:
This will be a single arm, prospective cohort study.

The names of the study intervention involved in this study is:

* Cone Beam Computed Tomography (CBCT)-guided electromagnetic navigational bronchoscopy (ENB) microwave ablation (MWA)
* A rapid on-site evaluation (ROSE) will be performed before the MWA to confirm that the lesion is malignant, this can lead to longer procedure time and time under anesthesia.

The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.

* Participants will receive the study intervention and will be followed for 30 days.
* It is expected that about 10 people will take part in this research study.

This research study is a Pilot Study, which is the first-time investigators are examining this intervention using a bronchoscopic approach for microwave ablation of solitary pulmonary nodules.

The U.S. Food and Drug Administration (FDA) has approved this intervention as a treatment option for this disease.

ELIGIBILITY:
Inclusion Criteria:

* Subject with Stage I - II primary lung cancer (Solitary nodules up to 3 cm) as defined by previous pathology or ROSE.
* Pathological proof of target nodule/tumor type and malignancy with specimen considered adequate per institutional laboratory standards
* Target nodule/tumor which can be accessed via navigational bronchoscopy and confirmed location with cone beam CT scan intra-operatively
* Resection/surgical candidate (lobectomy or greater)
* Participants must be at least 22 years old and able to provide consent

Exclusion Criteria:

* Subjects in whom flexible bronchoscopy is contraindicated
* Target nodule < 1.0 cm
* Prior radiation or neo adjuvant chemotherapy of the target nodule/tumor
* Any comorbidity that the investigator feels would interfere with the safety of the subject or the evaluation of study objectives
* Pacemaker, implantable cardioverter, or another electronic implantable device
* Patient cannot tolerate bronchoscopy
* Patients with coagulopathy
* Patients in other therapeutic lung cancer studies
* Subject is pregnant or breastfeeding
* COVID-19 positive patient at the time of procedure.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of Planned Ablations. | Day 1
  Feasibility of performing the procedure as planned in the enrolled patients. At least 9/10 of the planned ablations (90%) can be performed bronchoscopically according to the established protocol.
Pathological changes in the tumor tissue. | 4 weeks
  Pathological evaluation of the acute thermal effect produced by the AveCUre 16G-FMAP on targeted malignant solitary lung nodules will be described. The % necrosis, % viable tumor, and % stroma/inflammation present in the targeted nodules after ablation will be described.

SECONDARY OUTCOMES:
Histological changes in lung tissue outside the zone of predicted ablation. | 4 weeks
  A secondary analysis of the tissue surrounding the treated area will be performed. The % necrosis and of % stroma/inflammation will be described.
Immune-histochemical changes in the tumor tissue. | 4 weeks
  Immune-histochemical evaluation including TTF-1, Napsin-A, p40, or other immune-histochemical assessments will be performed if needed on a per case basis.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Beattie, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu

REFERENCES:
- [Derived] Beattie J, Parrish R, Ayasa L, Aranguren P, Uribe-Buritica FL, Lopez MN, Pineda CM, Cheng G, Senitko M, Abdelghani R, Magge A, Avendano CA, Kheir F, Swenson K, Parikh M, Wilson J, VanderLaan PA, Gangadharan S, Majid A. Safety and feasibility of bronchoscopic microwave ablation technology for peripheral lung cancer: a multi-center, prospective, single-arm study protocol. BMC Surg. 2025 Oct 24;25(1):497. doi: 10.1186/s12893-025-03230-y. PMID 41137055